CLINICAL TRIAL: NCT06354933
Title: Neurological Soft Signs in Neurodegenerative Dementias
Acronym: DemeNSS
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: DemeNSS (3785)
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease; Dementia With Lewy Bodies; Frontotemporal Dementia; Corticobasal Degeneration
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Frontotemporal Dementia; Corticobasal Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurodegenerative dementias: Subjects with either Alzheimer's disease, frontotemporal dementia, dementia with Lewy bodies or corticobasal syndrome
  Interventions: Diagnostic Test: Neurological Soft Signs
- Control: Subjects without dementia
  Interventions: Diagnostic Test: Neurological Soft Signs

INTERVENTIONS:
Diagnostic Test: Neurological Soft Signs — Neurological Soft Signs score according to the Heidelberg Manual

SUMMARY:
The goal of this observational study is to investigate the prevalence of Neurological Soft Signs (NSS) in various categories of dementia patients compared to matched controls. The main questions it aims to answer are:

* Does the prevalence of NSS significantly differ among patients with neurodegenerative dementias compared to controls?
* Are NSS associated with neuropsychiatric alterations in dementia patients?
* Do NSS correlate with cognitive screening tools?
* Do NSS increase over time in patients with neurodegenerative dementias?

Participants will undergo assessments including:

* Evaluation of NSS using the Heidelberg scale
* Neuropsychiatric assessments
* Cognitive screening using the Mini-Mental State Examination (MMSE) and Frontal Assessment Battery (FAB)

Researchers will compare dementia groups (Alzheimer's disease, Frontotemporal dementia, Corticobasal syndrome and Lewy body dementia) to controls to determine differences in NSS prevalence. Additionally, associations between NSS and neuropsychiatric symptoms, as well as cognitive performance, will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's Disease (AD), Frontotemporal Dementia (FTD), Corticobasal Syndrome (CBS), or probable Lewy Body Dementia (LBD) according to established clinical criteria.
* MMSE score greater than 10.
* Age and gender-matched controls without a history of neurological or psychiatric conditions.

Exclusion Criteria:

* Mixed dementia or vascular etiology.
* History of neurological or psychiatric conditions predating the dementia diagnosis.
* Substance or alcohol abuse history.
* Known comorbidities affecting neurological or psychiatric function.
* MMSE score less than or equal to 10.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include individuals diagnosed with Alzheimer's Disease (AD), Frontotemporal Dementia (FTD), Corticobasal Syndrome (CBS), or Lewy Body Dementia (LBD), along with age and gender-matched controls without dementia. Controls will be recruited from caregivers and companions of patients attending other neurological clinics. All participants will undergo thorough neurological and neuropsychiatric assessments to confirm eligibility and evaluate outcomes.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Difference in NSS | 0 days (baseline)
  Difference in Neurological Soft Signs according to the Heidelberg manual between neurodegenerative dementias and controls (range 0-48, higher scores indicate worse performance)

SECONDARY OUTCOMES:
Association between NSS and Neuropsychiatric Inventory (NPI) scores | 0 days (baseline)
  Correlation between NSS and NPI (range 0-144) (higher values indicate better correlation)
Correlation between NSS scores and cognitive function assessed by Mini-Mental State Examination (MMSE) | 0 days (baseline)
  Correlation between NSS and MMSE (range 0-30) (higher values indicate better correlation)
Correlation between NSS scores and cognitive function assessed by Frontal Assessment Battery (FAB) | 0 days (baseline)
  Correlation between NSS and FAB (range 0-18) (higher values indicate better correlation)
Longitudinal changes in NSS scores | 12 months
  Longitudinal differences in NSS scores in subjects with neurodegenerative dementia (range 0-48) (higher scores indicate worse performance)

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Tremolizzo, MD, PhD, Principal Investigator — University of Milano Bicocca
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided